CLINICAL TRIAL: NCT06175546
Title: Determination of Duration of Wearing Compression Hosiery Necessary to Reduce Subjective Symptoms of Chronic Venous Disease
Brief Title: Daily Duration of Compression Treatment in Patients With Symptomatic Chronic Venous Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CompTreatCVD
Record Dates: First submitted 2023-12-06; First posted 2023-12-19 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-11

CONDITIONS: Chronic Venous Insufficiency; Varicose Veins of Lower Limb
Keywords: Chronic venous disease; Compression treatment; Compression socks; Treatment duration; Regimen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression regimen 6-8 hours per day 4 weeks (Experimental): 40 participants. A physical examination and duplex ultrasound of the veins of the lower extremities are performed. It is suggested to wear the compression socks 6-8 hours a day for 4 weeks
  Interventions: Device: Compression socks
- Compression regimen 10-12 hours per day 4 weeks (Active Comparator): 40 participants. An physical examination and duplex ultrasound of the veins of the lower extremities are performed. It is suggested to wear the compression socks 10-12 hours a day for 4 weeks
  Interventions: Device: Compression socks

INTERVENTIONS:
Device: Compression socks — Wearing of compression sock in prescribed regimen

SUMMARY:
Aim of study is to investigate the optimal duration and daily regimen of compression treatment in patients with chronic venous disease

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic chronic venous disease
* C0-C4 according to CEAP-classification

Exclusion Criteria:

* C5-C6 according to CEAP-classification
* Intolerance to compression socks
* Patient's unwillingness to use compression socks
* Inability to use compression socks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Leg discomfort related to CVD measured with 10-cm visual analogue scale (VAS) | Day 0, Day 7, Day 14, Day 21, Day 28
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no discomfort"/"no pain" anchor and the patient's mark, providing a range of scores from 0-100.
  The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Quality of life (QoL) was measured by ChronIc Venous Insufficiency Quality of Life (CIVIQ-20) | Day 0, Day 28
  There are 20 questions in the CIVIQ-20, each with 5 possible answers (1 to 5), the minimum possible score being 20 and the maximum 100. In order to calculate the GIS, the difference between the final score and the minimum possible score is to be divided by the difference between the theoretical maximum and minimum scores (100-20=80), multiplied by 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov Russian National Research Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No